CLINICAL TRIAL: NCT01486095
Title: Comparison of Healing Responses After Treatment of Complex Bifurcation Lesions With a Dedicated Bifurcation Device (Axxess™ Drug Eluting Coronary Bifurcation Stent System + Biomatrix™ Drug Eluting Coronary Stent System Stents in the Distal Branches) Versus the Culotte Technique Using Xience Prime Everolimus-eluting Stents : an Optical Coherence Tomography (OCT) Analysis
Brief Title: COmplex BifuRcation Lesions: a Comparison Between the AXXESS Device and Culotte Stenting: an Optical Coherence Tomography (OCT) Study
Acronym: COBRA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Biosensors International (Other)
Responsible Party: Principal Investigator, Prof Dr Walter Desmet, Christophe Dubois, MD, PhD, Principal Investigator, University Hospital, Gasthuisberg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UH Leuven S53441
Record Dates: First submitted 2011-11-28; First posted 2011-12-06 (Estimated); Last update posted 2017-05-09 (Actual); Status verified 2017-05

CONDITIONS: True Coronary Bifurcation Lesions

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AXXESS + Biomatrix (Experimental): After mandatory predilatation, a self-expanding, conically shaped nickel-titanium AXXESS biolimus A9-eluting stent is placed at the level of the carina. The device is available in 3.0 and 3.5 mm calibre and 11 and 14 mm length. Depending on the lesion anatomy, additional Biomatrix™ Drug Eluting Coronary Stent Systems are placed distally if necessary. The procedure is completed with kissing balloon postdilatation using non-compliant balloons sized to the reference vessel diameter of the distal branches. Before this kissing balloon inflation, consecutive high pressure inflations should be performed in both branches.
  Interventions: Device: AXXESS + Biomatrix Biolimus Eluting stent
- Culotte technique: Xience V/Prime (Active Comparator): The culotte technique consists of stenting one of both branches of the bifurcation lesion first, and after balloon dilatation of the stent meshes, stenting the uncovered branch through the first stent and leaving the main vessel covered with two overlapped stents. The procedure is terminated by kissing balloon dilatation of both branches using non-compliant balloons sized to the reference vessel diameter of the distal branches. Before this kissing balloon inflation, consecutive high pressure inflations should be performed in both branches.
  Interventions: Device: Culotte technique with Xience V or Xience Prime stents

INTERVENTIONS:
Device: AXXESS + Biomatrix Biolimus Eluting stent — NAP
  Arms: AXXESS + Biomatrix
Device: Culotte technique with Xience V or Xience Prime stents — NAP
  Arms: Culotte technique: Xience V/Prime

SUMMARY:
Treatment of bifurcation lesions with drug-eluting stents (DES) (especially when a double stent technique is used) is associated with a higher risk for stent thrombosis. Different factors may play a role in the higher risk for stent thrombosis in bifurcation lesions. Possible mechanisms are delayed endothelialisation due to the action of the drug, coating polymers, or overlapping stent segments, incomplete stent apposition at specific sites in the bifurcation lesion and higher thrombogenicity due to turbulent flow at the bifurcation site. In human pathological data, the RUTSS (ratio of uncovered to total stent struts) appears to be the most powerful predictor of stent thrombosis.

This prospective study will assess the differences in stent strut coverage and stent strut apposition after complex bifurcation lesion treatment with the dedicated AXXESS Biolimus A9-eluting bifurcation stent at the bifurcation site and additional Biomatrix Biolimus A9-eluting stents in the distal main vessel and the side branch versus treatment with the culotte technique using the Xience Prime everolimus-eluting stents.

DETAILED DESCRIPTION:
BACKGROUND: There is an ongoing controversy over the efficacy and safety of different bifurcation stenting techniques. Critical considerations are the rate of restenosis at the side branch ostium, and completeness of healing at sites of overlap of stent struts, which may affect the risk of stent thrombosis.

AIMS: To compare vessel healing at 9 months using OCT imaging for two different treatment techniques for treating bifurcation lesions. Quantitative assessment of OCT images will be used to assess re-endothelialisation and quality of strut apposition to the vessel wall.

METHODS: Patients with true bifurcation lesions with involvement of a significant side branch requiring a stent will be randomly assigned to one of two treatment strategies. Group A will comprise 20 patients which will be treated with the Axxess™ Drug Eluting Coronary Bifurcation Stent System (Biosensors Europe SA) where additional Biomatrix™ Drug Eluting Coronary Stent Systems (Biosensors Europe SA) are implanted into the distal main branch (MB) and the side branch (SB) as required. Group B will consist of 20 patients which will be treated with the culotte technique using Xience Prime everolimus-eluting stents (Abbott-Vascular, US). Kissing balloon dilatation using non-compliant balloons will complete the index procedure in all cases. At 9 months, control angiography for all patients (with QCA using dedicated software) and OCT (of both main vessel and side branch) will be performed.

ENROLMENT PLAN:

Start: Third quarter of 2011 Enrolment period: ± 12 months Clinical follow-up: 5 years Angiographic and OCT results expected third quarter of 2013

ELIGIBILITY:
Inclusion Criteria:

1. Patient older than 18 years
2. The subject has stable or unstable angina pectoris, or a positive functional study for ischemia.
3. The subject is eligible for PCI, and is an acceptable candidate for coronary artery bypass surgery.
4. The subject is male, or if female, has no childbearing potential or has had a negative urine or serum pregnancy test within 7 days of the index procedure and has no intention to become pregnant within a year of the procedure.
5. The subject has signed the informed consent prior to the procedure, and agrees to comply with the follow up requirements.
6. Patients with a de novo and true coronary bifurcation lesion (Medina classification (1,1,1), (1,0,1) or (0,1,1)).
7. Coronary artery with proximal parent vessel reference diameter of 2.75 - 3.75 mm and a branch vessel diameter of ≥ 2.25 mm.
8. The lesion must be at least 50% diameter stenosis within either the MB or SB.
9. Regarding lesion length: lesion should be able to be covered by 2 Xience Prime stents in a Culotte technique, or by a combination of maximally 1 AXXESS and 2 Biomatrix™ Drug Eluting Coronary Stents.
10. The side branch ostium is located at least 12 mm from the left main coronary artery.
11. The angle between the sidebranch and the parent vessel is less than 70°.

Exclusion Criteria:

1. Left ventricular ejection fraction of < 30%
2. Impaired renal function (serum creatinine > 2.0 mg/dl)
3. Previous and/or planned brachytherapy of target vessel
4. Lesion of the left main trunk > 50%, unprotected
5. The target vessel contains intraluminal thrombus.
6. The target lesion shows angiographic evidence of moderate to severe calcification or tortuosity.
7. Known allergies to antiplatelet, anticoagulation therapy, contrast media, everolimus or biolimus, stainless steel, cobalt, chromium, nickel or titanium
8. Pregnant and/or breast-feeding females or females who intend to become pregnant (pregnancy test required)
9. Patients with a life expectancy of less than one year
10. Patient currently enrolled in other investigational device or drug trial
11. Patient not able or willing to adhere to follow-up visits
12. Patients who intend to have a major surgical intervention within 6 months of enrolment in the study.
13. Patients who previously participated in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-11-29; Primary Completion 2013-12 (Actual); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint | 9 months
  Percent uncovered to total stent struts at 9 months, assessed with OCT, in two different bifurcation stenting techniques

SECONDARY OUTCOMES:
Secondary endpoint : stent strut coverage per segment with OCT | 9 months
  - Percent uncovered to total stent struts at 9 months per analyzed bifurcation segment (proximal MB, carina, distal MB, SB)
Secondary endpoint: stent strut apposition with OCT | 9 months
  - Percent malapposed to total stent struts at 9 months post procedure, both overall and per bifurcation segment
Secondary endpoint: clusters of malapposition with OCT | 9 months
  - Number of clusters of malapposition, overall and per bifurcation segment. Per cluster, the number of malapposed struts, the area (mm²), the volume (mm³) and the arc (degrees) of malapposition will be assessed.
Secondary endpoint: Tissue strut thickness with OCT | 9 months
  - Tissue strut thickness at 9 months per bifurcation segment (µm)
Secondary endpoint: neointimal hyperplasia volume | 9 months
  - Neointimal hyperplasia: absolute and percent volume of intimal hyperplasia at 9 months post procedure (mm³)
Secondary endpoint: late luminal loss (angiography) | 9 months
  - Late Lumen Loss (in-stent) at 9 months
Secondary endpoint: in-segment late luminal loss (angiography) | 9 months
  - In-segment Late Lumen Loss at 9 months (including stent + 5mm proximal and distal)
Secondary endpoint: binary restenosis (angiography) | 9 months
  - Binary in-stent restenosis at 9 months
Secondary endpoint: binary in-segment restenosis (angiography) | 9 months
  - Binary in-segment restenosis at 9 months (including stent + 5mm proximal and distal)
Secondary endpoint: minimal lumen diameter (angiography) | 9 months
  - Minimal Lumen Diameter (MLD), in-stent and in-segment at 9 months
Secondary endpoints: clinical: MACE | 1, 8 and 12 months and annually for 5 years from the procedure date
  - Cumulative MACE rate (cardiac death, Q- or non-Q-wave MI, or clinically driven TLR) at 1, 8 and 12 months and annually for 5 years from the procedure date.
Secondary endpoints: clinical: components of MACE: cardiac death | 1, 8 and 12 months and annually for 5 years from the procedure date
  - Cumulative components of MACE: cardiac death at 1, 8 and 12 months and annually for 5 years from the procedure date.
Secondary endpoints: clinical: components of MACE: Q- or non-Q-wave myocardial infarction | 1, 8 and 12 months and annually for 5 years from the procedure date
  - Cumulative components of MACE :Q- or non-Q-wave MI at 1, 8 and 12 months and annually for 5 years from the procedure date.
Secondary endpoints: clinical: components of MACE: clinically driven target lesion revascularization (TLR) | 1, 8 and 12 months and annually for 5 years from the procedure date
  - Cumulative components of MACE : clinically driven TLR at 1, 8 and 12 months and annually for 5 years from the procedure date.
Secondary endpoint: Stent thrombosis | 24h, 1 month, 12 months and yearly thereafter (up to 5y)
  - Stent thrombosis at at 24h, 1 month, 12 months and yearly thereafter (up to 5y)
Secondary endpoint: Target vessel revascularization | 1, 8, 12 months and yearly thereafter (up to 5y)
  - Target vessel revascularisation (TVR) at at 1, 8, 12 months and yearly thereafter (up to 5y)
Secondary endpoint: all-cause death | 1, 8, 12 months and yearly thereafter (up to 5y)
  - All-cause death at 1, 8, 12 months and yearly thereafter (up to 5y)
Secondary endpoint: non-target revascularization | 1, 8, 12 months and yearly thereafter (up to 5y)
  non-Target vessel revascularization at 1, 8, 12 months and yearly thereafter (up to 5y)
Secondary endpoint: any coronary revascularization | 1, 8, 12 months and yearly thereafter (up to 5y)
  Any coronary revascularization 1, 8, 12 months and yearly thereafter (up to 5y)
Secondary endpoint: device success | Immediately after initial treatment of the study lesion
  - Device success, defined as achievement of a final residual diameter stenosis of <30% measured by QCA.
Secondary endpoint: lesion treatment success | Immediately after initial treatment of the study lesion
  - Lesion treatment success, defined as <30% residual stenosis in the MB and <50% in the SB measured by QCA by any treatment.
Secondary endpoint: procedure success | 24h after treatment of the target lesion
  - Procedure success, defined as lesion success without the occurrence of MACE during the hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe L Dubois, MD, PhD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven
Locations (2):
- Belgium (2):
  - ZOL Genk, Genk
  - UH Leuven, Leuven